CLINICAL TRIAL: NCT06715631
Title: Human Factors Validation Testing of the Wandercraft Personal Exoskeleton
Acronym: ExoUser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP010
Record Dates: First submitted 2024-11-18; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries; Tetraplegia; Paraplegia
Keywords: Spinal Cord Injuries; Robotics; Community use; Hands-free exoskeleton; Overground exoskeleton; Walking; Self-balancing
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paraplegia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hands-free exoskeleton (Experimental)
  Interventions: Device: Hands-free exoskeleton

INTERVENTIONS:
Device: Hands-free exoskeleton — Before the simulated-use test, the SCI user and his/her companion must attend five training sessions provided by a Wandercraft certified trainer. Training will be composed by a theoretical part including presentation and description of the personal exoskeleton and its use modes and a hands-on practice. Each session lasts between 1 to 2 hours, varying according to the user's learning pace and tolerance. The training program is representative of the intended training for the end product.

SUMMARY:
The goal of this interventional, national, prospective, open and monocentric study is to demonstrate that a personal exoskeleton can be used by the intended users without serious use errors or problems, for the intended uses and under the expected use conditions.

DETAILED DESCRIPTION:
The Atalante X exoskeleton, Wandercraft's first-generation hands-free, self-balancing device covered by an EC certificate and cleared by the FDA, was primarily utilized in rehabilitation institutions. However, recognizing the potential benefits of self-balancing exoskeleton technology in home settings for individuals with paraplegia and tetraplegia, Wandercraft developed a personal exoskeleton designed for home and community use.

The scope of this protocol is to validate all the critical tasks performed by the intended SCI users and companions of the device, according to IEC 62366-1(2020) and the FDA Guidance "Applying human Factors and Usability Engineering to Medical Devices.

Up to 14 participants will be recruited and will include:

* SCI users: adult patients with motor complete or incomplete SCI with a clinical presentation of a neurological level at or above T6,
* Companions: adult individuals in charge of assisting the patient during the use of the device.

Both the SCI user and their companion must complete a joint certification program to ensure safe and effective use of the device. The program is provided by a Wandercraft certified trainer and consists of five sessions spread over a maximum period of two months. These sessions include both theoretical presentations on the exoskeleton and practical hands-on training. As a precautionary measure in this usability study, a safety rail will be used to secure the user but it will not be part of the final product.

Usability will be assessed by:

1. IFU questionnaire,
2. Simulated tasks test,
3. Final debriefing.

ELIGIBILITY:
SCI user inclusion criteria:

* Any gender, age 18 years old or older.
* Motor complete or incomplete SCI with a clinical presentation of a neurological level at or above T6.
* Has been released from acute inpatient care following their SCI.
* Able and willing to attend 6 one-to-two-hour sessions of training.
* Able to read, understand, and provide informed consent.
* Patients affiliated to a social security system.

SCI user exclusion criteria:

* Any neurological injury other than spinal cord injury (SCI), except where such injury does not result in physical disability
* Progressive condition that would be expected to result in changing neurological status.
* Severe concurrent medical disease, illness or condition judged to be contraindicated by the site physician.
* Unhealed or unstable traumatic or high impact lower extremity fracture of any duration that is, in the clinical judgement of the study physician, exclusionary for standing and walking.
* Individual with history of osteoporotic fracture and / or pathology or treatment causing secondary osteoporosis.
* Untreatable severe spasticity judged to be contraindicated by the site physician.
* Untreated/uncontrolled hypertension as judged to be contraindicated by the site physician.
* Unresolved orthostatic hypotension as judged to be contraindicated by the site physician.
* History of uncontrolled autonomic dysreflexia.
* Presence of colostomy and/or urostomy.
* Ventilator use at the time of exoskeleton use.
* Presence of life supporting device (e.g., pacemaker).
* Open or unhealed skin pressure sores, abrasions, or bruises at any of the contact points of the exoskeleton.
* Morphological contraindications to the use of the device.
* Uncorrectable leg length discrepancy over 2 cm (about 0.79 in) when using additional correction tools.
* Individuals with functional and/or cognitive impairments that prevent them from effectively operating the device using a hand control interface.
* Improper fitting in the device.
* Psychopathology documentation in the medical record that may conflict with study objectives.
* Pregnancy or women who plan to become pregnant during the study period.
* Concurrent participation in another interventional trial.
* Patient under legal protection.

Companion inclusion criteria:

* Any gender, age 18 years or older.
* Able and willing to attend 6 one-to-two-hour sessions of training.
* Able to read, understand and provide informed consent.

Companion exclusion criteria:

* Inability to communicate with an assistant due to cognitive or language disorders.
* Any disease, concomitant injury, or condition that interferes with the performance or interpretation of the protocol- specified assessments.
* Insufficient strength and performance capability, evidenced by the ability to hold and retain the device in case of unbalance/fall.
* Presence of life supporting device (e.g., pacemaker).
* Concurrent participation in another interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
SCI user and companion performance when carrying out tasks that are critical tasks | At session 6, after an average of 7.5 hours of training.
  The acceptance criterion for this test is 100% of the trained SCI users and trained companions are able to perform each of the critical task successfully during a simulated-use test.

SECONDARY OUTCOMES:
Use errors, close calls, and use difficulties | At session 6, after an average of 7.5 hours of training.
  Collection of observed use errors, close calls, and use difficulties and identification of critical issues during a simulated-use test - no passing criteria.
SCI user and companion general performance when carrying non-critical tasks | At session 6, after an average of 7.5 hours of training.
  The acceptance criterion for this test is 90% of the trained SCI users and trained companions are able to perform each of the non-critical task successfully during a simulated-use test.
Readability and clarity of Instructions for Use (IFU) | At session 5, after an average of 6 hours of training.
  The acceptance criteria for this test is 100% of the SCI users and companions are able to answer to the critical task questions of the IFU questionnaire correctly and 90% are able to answer to the non-critical task questions correctly.
SCI user and companion opinion on the accompanying documents and training | At session 6, after an average of 7.5 hours of training.
  The acceptance criterion for this test is 90% of the trained SCI users and trained companion rate the accompanying documents and training 3 or higher using 5-level Likert scale (1 inadequate, 2 barely adequate, 3 neither adequate nor inadequate, 4 adequate, 5 satisfactory).

OTHER OUTCOMES:
SCI user and companion satisfaction and comfort | At session 6, after an average of 7.5 hours of training.
  Evaluation of the SCI user and companion satisfaction and comfort on the user interfaces and use modes using 5-level Likert scales. Gather feedback on recommended changes through open-ended questions - no passing criteria.
Usability of donning and doffing | At session 6, after an average of 7.5 hours of training.
  Measurement of the time required for donning and doffing during a simulated-use test - no passing criteria.
Functional test with the exoskeleton | At session 6, after an average of 7.5 hours of training.
  Evaluation of the SCI user performance (i.e., success and timing) during a Timed Up andGo (TUG) test with the exoskeleton - no passing criteria.
SCI user fitting within the device | Through study completion, an average of 9 hours of training and assessment.
  Assessment of the SCI user skin in the areas of contact with the exoskeleton - no passing criterion.
Frequency and type of exoskeleton imbalances corrected by the safety rail and by the companion | Through study completion, an average of 9 hours of training and assessment.
  Collection of data regarding the frequency and type of exoskeleton imbalances corrected by the safety rail and by the companion - no passing criteria.
Assistance provided by the companion during device use | At session 6, after an average of 7.5 hours of training.
  Evaluation of the level of assistance provided by the companion during the execution of the functional test and donning and doffing - no passing criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sauvagnac, MD, Principal Investigator — Wandercraft
Locations (1):
- Wandercraft, Paris, France